CLINICAL TRIAL: NCT07166380
Title: An Open-label, Blinded Ib/IIa Study Investigating the Treatment of Acute Large Hemispheric Infarction by Transcranial Bone Marrow Injection of RK-4 Injection
Brief Title: RK-4 Intracalvariosseous Injection in Treatment of Acute Large Hemispheric Infarction
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Collaborators: Fuzhou Neurodawn Rongkang Pharmaceutical Co., Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RK-4-LC-01
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Transcranial Bone Marrow Injection; RK-4; Acute Large Hemispheric Infarction; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RK-4 injection (Experimental): patients will take drug RK-4 (1 mg or 2 mg or 4 mg) by transcranial bone marrow injection once daily for consecutive 3 days.
  Interventions: Drug: RK-4 injection

INTERVENTIONS:
Drug: RK-4 injection — patients with LHI will take drug RK-4 (1 mg or 2 mg or 4 mg) by transcranial bone marrow injection once daily for consecutive 3 days.

SUMMARY:
An open-label, blinded Ib/IIa study investigating the treatment of acute large hemispheric infarction by transcranial bone marrow injection of RK-4 injection

For subjects with acute large hemispheric infarction who are contraindicated to vascular recanalization or have poor response to vascular recanalization therapy, the safety, tolerability, and PK characteristics of RK-4 injection injected into the brain cell marrow through the cranial bone marrow will be preliminarily evaluated, and the efficacy will be preliminarily explored. The main questions it aims to answer are:

* If drug RK-4 is safe and tolerate in the patients with LHI?
* What the pharmacokinetic profiles of RK-4 injection injected into the brain cell marrow through the cranial bone marrow?
* The efficacy of RK-4 injection injected into the brain cell marrow through the cranial bone marrow Researchers will analyze data from different groups, includes low dose group (1mg，QD), medium dose group(2mg，QD), high dose group(4mg，QD), to see If drug RK-4 is safe and tolerate in the patients with LHI and the pharmacokinetic profiles and efficacy of RK-4 injection injected into the brain cell marrow through the cranial bone marrow.

Participants will:

* Take drug RK-4 (1 mg or 2 mg or 4 mg) by transcranial bone marrow injection once daily for consecutive 3 days.
* Truthfully provide medical history and "previous participation in clinical trials" and a statement of no history of mental disorders.
* Take the drug at the specified time every day according to the dosage prescribed by the doctor
* Receive the investigational drug as instructed by the doctor and visiting as required
* Tell the investigators about any medications (including chemicals, biological drugs, proprietary Chinese medicines, etc.) and related treatments you take during the study
* unpermitted stop the investigational drug yourself at the end of the study or when you decide to withdraw from the study, you need to stop the investigational drug as directed by your doctor to ensure your safety
* take reasonable contraception actions
* unallowed to use unmarketed drugs or other clinical trial drugs during the study

ELIGIBILITY:
Inclusion Criteria:

1. 18≤ age < 81 years old, gender is not limited;
2. The modified Rankin score (mRS) score ≤ 1 point before the onset of stroke;
3. Administration can be completed within 24 hours after the onset of symptoms and signs of neurological deficit (for subjects with stroke after waking up or stroke without witnesses, the last normal time of symptom onset is the time of symptom onset);
4. Clinical symptoms, signs and imaging diagnosed as cerebral infarction in the middle cerebral artery blood supply area, and the following characteristics are met:

   1. 16≤NIHSS score ≤32 points, sum of the fifth upper limb and sixth lower limb scores≥6;
   2. Imaging suggests the core area of infarction: cerebral blood flow (CBF) in electronic computed scan perfusion imaging (CTP) < 30% volume or apparent diffusion coefficient (ADC) value in magnetic resonance imaging (MRI) diffusion-weighted imaging (DWI) sequence < 70-300ml of 620×10-6mm2/s lesion volume or ASPECTS score of 0-6 points. Priority is given to CTP test results. If both CTP and DWI are completed during the screening period and the examination results are inconsistent, the investigator needs to take all information (scanning time, imaging method for optimal response infarct size, etc.) into account and then make a reasonable judgment and record that; ASPECTS scores can be based on CTP or MRI, but CTP is preferred.
5. If vascular reperfusion therapy is performed, the treatment is not effective and the following conditions are met:

   1. Extended thrombolytic grading (eTICI) = 2a;
   2. NIHSS score did not improve or progressed after vascular reperfusion treatment and the total score was still ≤ 32 points.

   Note: A decrease of 1 point or more is an improvement, and an increase of 1 point or more is progress.
6. Subjects or their legal representatives voluntarily sign the informed consent form.

Exclusion Criteria:

-

Those who meet one of the following items at screening cannot be enrolled:

1. Concurrent cerebrovascular disease meets one of the following conditions:

   1. Combined with acute cerebral hemorrhage and subarachnoid hemorrhage;
   2. Combined with acute posterior circulation cerebral infarction, or severe posterior circulation vascular stenosis (>70%);
   3. Imaging suggests bilateral involvement of the cerebral infarction area;
   4. The cause has been diagnosed by TOAST typing before screening, and other etiologies such as intracranial artery dissection, vasculitis, and moyamoya disease have been identified
2. Hemorrhage transformation in the infarct area, the hematoma area ≥ 30% of the infarcted area, and has an obvious mass occupancy effect;
3. Presence of clinical signs of cerebral herniation, e.g., unilateral or bilateral pupil dilation, fixation; Cerebral edema-related loss of consciousness (NIHSS 1a>2 points), or other brainstem reflex loss judged by the investigator caused by cerebral edema or cerebral herniation formation; or other unstable signs of vital signs that are difficult to control;
4. Planned cranial decompression flap decompression at screening;
5. Refractory hypertension (systolic blood pressure >200mmHg or diastolic blood >110mmHg) or hypotension (systolic blood pressure <70mmHg or diastolic blood pressure <50mmHg) that is difficult to control with medication;
6. Abnormal blood glucose (random venous blood glucose < 2.8mmol/L or >23mmol/L);
7. Obvious abnormal liver function indicators or obvious abnormal renal function indicators; Note: Obvious abnormalities in liver function indicators refer to serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN); Significant abnormal renal function measures are defined as eGFR less than 60 mL/min/1.73 m² (eGFR is calculated using the CKD-EPI formula).
8. Acute ST-segment elevation myocardial infarction (MI), and/or acute decompensated heart failure (according to New York College of Cardiology (NYHA) cardiac function class III and IV) within the past 3 months];
9. Contraindications to transcranial bone marrow administration, such as skull fracture, skull infection, subdural/external hematoma, subscalp hematoma, scalp skin or subcutaneous infection, cranial plate obstruction in the past 3 months, etc.;
10. Bleeding tendency that is not conducive to operation in the opinion of the investigator, including but not limited to: platelet count <100×109/L, presence of coagulation dysfunction diseases such as hemophilia, etc.;
11. Presence of severe or very severe anemia (hemoglobin < 60 g/L);
12. Combined with severe respiratory diseases (severe chronic obstructive pulmonary disease, respiratory failure, etc.) that need to be corrected by endotracheal intubation, tracheostomy or ventilator;
13. Subjects have severe local or systemic infections within 3 days before screening, including but not limited to severe local symptoms due to infection, such as suppuration, severe pain, tissue necrosis, or clear systemic infection-related symptoms, such as rapid onset of high fever (>38.5°C), rapid heart rate, chills, impaired consciousness, dyspnea, shock, etc. caused by infection;
14. Diagnosed serious CNS degenerative diseases, such as Alzheimer's disease (AD), Parkinson's disease (PD) and severe dementia caused by various reasons or mental system diseases (such as schizophrenia, depression, etc.);
15. Previously diagnosed with severe systemic disease, with an expected survival of < 90 days;
16. Known allergy to any component of the treatment drug and contrast agent during the study process;
17. Subjects who are pregnant, lactating, or have possible pregnancy and plan to become pregnant;
18. Subjects are unable to comply with the study protocol or follow-up requirements;
19. Those who have participated in any other interventional clinical trial within 3 months before screening, or are currently participating in any other clinical trial;
20. The investigator believes that he is not suitable to participate in this clinical study.

After enrollment, if the subject is found to have violated the enrollment criteria or met the exclusion criteria; such as the age is found to be greater than or equal to 81 years old or malignant tumors or other aspects that do not meet the inclusion criteria, the investigator can judge whether it is suitable to continue to participate in the study based on the risks and benefits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of RK-4 in patients with LHI by incidence of subject getting abnormal results of physical examinations after treatment. | Day1 ~Day 14
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation
Evaluate the tolerability of RK-4 in patients with LHI by incidence of subject getting abnormal results of physical examinations after treatment. | Day1 ~Day 14
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation
Evaluate the safety of RK-4 in patients with LHI by incidence of subject getting abnormal results of vital signs after treatment. | Day1 ~Day 14
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(blood pressure, respiration, pulse, body temperature） will be assessed by according equipments.(electronic sphygmomanometer，thermometer).
Evaluate the tolerability of RK-4 in patients with LHI by incidence of subject getting abnormal results of vital signs after treatment. | Day1 ~Day 14
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(blood pressure, respiration, pulse, body temperature） will be assessed by according equipments.(electronic sphygmomanometer，thermometer).
Evaluate the safety of RK-4 in patients with LHI by incidence of subject getting abnormal results of 12-lead ECG after treatment. | Day1 ~Day 14
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Evaluate the tolerability of RK-4 in patients with LHI by incidence of subject getting abnormal results of 12-lead ECG after treatment. | Day1 ~Day 14
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Evaluate the safety of RK-4 in patients with LHI by incidence of subject getting abnormal results of laboratory tests after treatment. | Day1 ~Day 14
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Evaluate the tolerability of RK-4 in patients with LHI by incidence of subject getting abnormal results of laboratory tests after treatment. | Day1 ~Day 14
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.
Evaluate the safety of RK-4 in patients with LHI by rates of adverse events after treatment. | Day1 ~Day 14
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment.
  The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of CTCAE 5.0.
  The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.
Evaluate the tolerability of RK-4 in patients with LHI by rates of adverse events after treatment. | Day1 ~Day 14
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment.
  The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of CTCAE 5.0.
  The relevance evaluation is divided into 5 grades: 1-certainly related; 2- probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.

SECONDARY OUTCOMES:
Evaluate the Cmax of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin | Day1 ~Day 5
  Maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the AUC 0-t of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin. | Day1 ~Day 5
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration.
  Calculated according to linearity trapezoidal rule:
  AUC (i, i+1) = (Ti+1-Ti) (Ci+Ci+1) /2, and AUC0-t is the sum of all AUC (i, i + 1)
Evaluate the AUC 0-∞ of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin. | Day1 ~Day 5
  Area under the concentration-time curve from time 0 to infinity (extrapolated). AUC 0-∞ =AUC 0-t + Ct/λz (Ct is the last measured plasma concentration).
Evaluate the Tmax of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin. | Day1 ~Day 5
  Time to reach maximum observed plasma concentration. It was obtained directly from the measured plasma concentration-time data.
Evaluate the t1/2 of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin. | Day1 ~Day 5
  Terminal elimination half-life. t1/2 = ln2/λ
Evaluate the λz of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin. | Day1 ~Day 5
  Terminal-phase elimination rate constant, slope of curves terminal segment at semi-log concentration-time curve calculated by linear regression.
Evaluate the AUC_%Extrap of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin | Day1 ~Day 5
  The percentage of the AUC0-inf that has been extrapolated. AUC_%Extrap = [(AUC0-∞-AUC0-t)/AUC0-∞] × 100%
Evaluate the Vz of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin | Day1 ~Day 5
  Volume of distribution. Vz = Div/AUC0-∞/λz
Evaluate the CL of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin. | Day1 ~Day 5
  Total body clearance. CLz = Div /AUC0-∞
Evaluate the MRT 0-t of single ascending doses of RK-4 in patients with LHI by venous blood and Phoenix WinNonlin. | Day1 ~Day 5
  Mean residence time within the time from time zero to the lowest testing plasma concentration. MRT0-t = AUMC0-t/AUC0-t
Evaluate the efficacy of RK-4 in patients with LHI by the proportion of NIHSS score improvement of ≥8 points from baseline | Day 14
  National Institute of Health stroke scale(NIHSS) is a scale used to assess neurological function. it contains 15 items, with a total score of 0-42. The lower the score is, the better neurological function the patient has.
Evaluate the efficacy of RK-4 in patients with LHI by the proportion of NIHSS score improvement of ≥4 points from baseline | Day 14
  National Institute of Health stroke scale(NIHSS) is a scale used to assess neurological function. it contains 15 items, with a total score of 0-42. The lower the score is, the better neurological function the patient has.
Evaluate the efficacy of RK-4 in patients with LHI by the change of NIHSS score from baseline | Day4, Day8, Day14
  National Institute of Health stroke scale(NIHSS) is a scale used to assess neurological function. it contains 15 items, with a total score of 0-42. The lower the score is, the better neurological function the patient has.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TianTan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No